CLINICAL TRIAL: NCT05403905
Title: A Cohort Study of Non-surgical Treatment and Exercise Rehabilitation in Patients -Chinese Population-based Cohort
Brief Title: A Cohort Study of Non-surgical Treatment and Exercise Rehabilitation in Patients With Anterior Cruciate Ligament Rupture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006761-M2022073
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Anterior Cruciate Ligament Rupture; Osteoarthritis, Knee
Keywords: Anterior cruciate ligament (ACL); OA; non-surgical treatment; rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Osteoarthritis, Knee | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: The patients who were diagnosed with complete rupture of the ACL in the outpatient department of Peking University Third Hospital, the sports medicine doctor explained in detail (1) the way of conservative treatment, (2) the ruptured anterior cruciate ligament has the possibility of healing after fixation and (3) Willing to join the cohort study after enrollment. There were 60 subjects in the non-surgical treatment group and 60 in the surgical treatment group, for a total of 120 subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-surgical treatment (Experimental): The patient who was diagnosed with complete rupture of the ACL in the Institute of Sports Medicine of the Third Hospital of Peking University was informed by the doctor that there is a chance that the ACL may grow back after 6 weeks of strict bracing.
  Interventions: Procedure: non surgical treatment
- surgical treatment (Active Comparator): The patient who was diagnosed with complete rupture of the ACL in the Institute of Sports Medicine of the Third Hospital of Peking University was informed by the doctor that there is a chance that after 6 weeks of strict brace immobilization, the ACL may grow back without surgery. However, the choice was still made for immediate ACL reconstruction.
  This group of patients underwent anterior cruciate ligament reconstruction surgery in the Third Hospital of Peking University.
  Interventions: Procedure: surgical treatment

INTERVENTIONS:
Procedure: non surgical treatment — Conservative treatment is required to use a curved splint for 6 weeks to keep the feet on the ground, bathing and sleeping without loosening the utensils and taking no steroids during the period. Physical examination and magnetic resonance imaging were performed after 6 weeks. If laxity remained unsatisfactory, the outcome was recorded as failure and surgery was changed.
  Arms: non-surgical treatment
Procedure: surgical treatment — The patient underwent knee arthroscopic anterior cruciate ligament surgery at the Institute of Sports Medicine of the Third Hospital of Peking University. The surgical methods were all anatomical single-bundle.
  Arms: surgical treatment

SUMMARY:
This clinical trial compared the prognosis of surgical and non-surgical treatment in patients with complete anterior cruciate ligament rupture

DETAILED DESCRIPTION:
Anterior cruciate ligament injury is a common neuromuscular injury to the knee joint. The incidence rate is gradually increasing. There are 400,000 ACL reconstruction operations in the United States every year. The population of my country is equivalent to 4.3 times that of the United States. The potential economic burden of cruciate ligament reconstruction surgery on the country cannot be ignored. Anterior cruciate ligament reconstruction is seen as an effective treatment for this disease, avoiding secondary meniscus damage and knee degeneration, but the failure rate is still as high as 20%. In addition, problems such as poor bending angle caused by postoperative adhesions that may occur after surgery, atrophy of the quadriceps muscle of the patient's affected leg, and overstrain of the healthy leg caused by psychological factors may affect the quality of life after surgery. Reasons that prevent return to sports. The use of conservative treatment instead of surgery after recent ACL injury has received high attention, and a large number of RCTs have compared the benefits of surgery and conservative treatment.

Some reviews pointed out that the clinical outcomes of surgical treatment and conservative treatment are not much different, and even questioned the prognosis after anterior cruciate ligament reconstruction. Individual differentiated treatment is necessary.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 8-45 years old 2) Complete rupture of unilateral anterior cruciate ligament (ACL) (with/without partial meniscus tear) 3) The history of ACL injury should not be more than 2 months before enrollment 4) Complete rupture of the ACL as determined by clinical examination and MRI 5) Activity level scale 5-9 (Tegner activity score) 6) Degeneration of knee joint <KL II degree, intraoperative cartilage injury < ICRS III degree.

  7) The reason for the rupture of the anterior cruciate ligament is sports trauma.

  8) Complete rupture of the ACL meets the MRI indications: (1) The signal changes, deforms, and thickens on imaging, and is completely broken but not separated; (2) There is no sagging and separation of the broken ends; (3) The synovial image is continuous.

  9) The physical examination of complete ACL rupture meets the following indications: (1) Lachman (-) or ADT (-) has one of them; (2) or both are slightly loose, and the slack is not more than 10mm; (3) vertical Leg position ADT (-) or slack <5mm.

Exclusion Criteria:

* 1) Used in the previous 12 months 1. Intra-articular injection 2. Physical therapy 2) Those who broke again after surgery and underwent knee surgery in other hospitals 3) Previous knee surgery (except diagnostic arthroscopy) 4) Active infection of the knee joint within the past 12 months 5) Informed consent cannot be given 6) History of knee gout 7) Include one or more of the following knee-related injuries: 8) Unstable meniscus tears requiring repair or post-operative changes in rehabilitation Bicompartmental wide meniscectomy Total collateral ligament rupture full thickness cartilage lesions 9) History of rheumatoid arthritis or similar rheumatic diseases 10) The discovery of rheumatoid arthritis, rheumatoid arthritis pigment villonodular synovitis and other joint diseases during the postoperative follow-up period may impair the ability to participate in the study 11) Unable to speak/understand the research content, lack of autonomy, unable to walk, or unable to participate in follow-up 12) Participate in any drug trials during and after the disease 13) Any other medical condition that considers the longest survival time to be less than 2 years 14) Immunodeficiency or HIV positive 15) Illegal drug use or chronic alcoholism or total daily alcohol intake > 50 g/d 16) Pregnancy/planning pregnancy 17) There are contraindications such as current or previous history of neurological disease, cerebrovascular and serious cardiovascular disease, including coronary heart disease (angina pectoris, myocardial infarction, coronary angiogenesis process or abnormal electrocardiogram Q wave appearance (ECG)), Stroke (ischemic or hemorrhagic, including transient ischemic attack), peripheral arterial disease diagnosed by angiography 18) No imaging diagnosis 19) History of deep vein thrombosis (DVT) or blood system 20) There is a systemic disease that affects physical function, or there is any other condition or treatment that prevents the completion of the trial, including patients with metal devices or movement disorders

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form 2000 | At 6 months after intervention.
  Patients will be asked to fill out the IKDC2000 score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.The role of IKDC2000 is not only to compare the prognosis of the knee joint between the surgical group and the non-surgical group, but also to the normal population we mentioned in the article according to The International Knee Documentation Committee Subjective Knee Evaluation Form Normative Data Allen F. Anderson,*† AJSM The IKDC2000 values of different genders and ages were used to judge whether the two groups of patients reached the standard of normal people after surgery.
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form 2000 | At 12 months after intervention.
  Patients will be asked to fill out the IKDC2000 score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.The role of IKDC2000 is not only to compare the prognosis of the knee joint between the surgical group and the non-surgical group, but also to the normal population we mentioned in the article according to The International Knee Documentation Committee Subjective Knee Evaluation Form Normative Data Allen F. Anderson,*† AJSM The IKDC2000 values of different genders and ages were used to judge whether the two groups of patients reached the standard of normal people after surgery.
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation | At 24 months after intervention.
  Patients will be asked to fill out the IKDC2000 score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.The role of IKDC2000 is not only to compare the prognosis of the knee joint between the surgical group and the non-surgical group, but also to the normal population we mentioned in the article according to The International Knee Documentation Committee Subjective Knee Evaluation Form Normative Data Allen F. Anderson,*† AJSM The IKDC2000 values of different genders and ages were used to judge whether the two groups of patients reached the standard of normal people after surgery.
Quadriceps strength | At 24months after intervention.
  Side to side quadriceps strength assessed by Biodex arthrometer test
Knee laxity （physical exam） | At 24months after intervention.
  The side to side knee joint laxity of patients after anterior cruciate ligament surgery can be divided into four grades: grade A: -1~2mm(0+), grade B: 3~5mm (1+), grade C: 6~10mm (2+) and D Grade: >10mm(3+) assessed by Lachman test of physical examination.
Knee laxity （KT-2000 arthrometer） | At 24months after intervention.
  The knee laxity test of the forward KT-2000 measured knee laxity at pressures of 132Nt, 88Nt, 66Nt, and 44Nt, respectively, while the back-pushing KT-2000 was measured at -132NT, 88Nt, 66Nt, and -44Nt. The foward-pushing KT-2000 asessed side-to-side can be stratified into five levels are (A) < - 1 mm, (B) - 1 to 1 mm, (C) 1-3 mm, (D) 3-5 mm and (E) > 5 mm.
  The back-pushing KT-2000 is also divided into side to side differences as (A) < - 2 mm, (B) - 2 to - 0.5 mm, (C) - 0.5 to 0.5 mm, (D) 0.5-1 mm and ( E) > 1 mm.
Magnetic resonance imaging (MRI) | At 24months after intervention.
  Magnetic resonance imaging was used to compare lateral comparisons of ligament healing and ACL graft healing after conservative treatment, meniscal damage and knee cartilage damage after intervention.

SECONDARY OUTCOMES:
Gender | At baseline.
  Measuring whether gender is a risk factor for anterior cruciate ligament reconstruction failure.
Age | At baseline
  Measuring whether age is a risk factor for anterior cruciate ligament reconstruction failure
BMI | At baseline
  Weight and height will be combined to report BMI in kg/m^2. Measuring whether bmi is a risk factor for anterior cruciate ligament reconstruction failure
Single-Legged Hop Test | At 6 months after intervention.
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the single hop for distance.
Single-Legged Hop Test | At 12 months after intervention.
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the single hop for distance.
Single-Legged Hop Test | At 24 months after intervention.
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the single hop for distance.
Triple hop test | At 6 months after intervention.
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the triple hop for distance.
Triple hop test | At 12 months after intervention.
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the triple hop for distance.
Triple hop test | At 24 months after intervention.
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the triple hop for distance.
Cross hop test | At 6 months after intervention.
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the cross hop for distance.
Cross hop test | At 12 months after intervention.
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the cross hop for distance.
Cross hop test | At 24 months after intervention.
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the cross hop for distance.
6-m hop test | At 6 months after intervention.
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the 6-meter hop for time.
6-m hop test | At 12 months after intervention.
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the 6-meter hop for time.
6-m hop test | At 24 months after intervention.
  The patients will perform three submaximal trial repetitions for familiarisation, after which three maximum effort trials are recorded. The uninvolved leg will test first at both inclusion sites. Record the 6-meter hop for time.
Knee Outcome Survey Activities of Daily Living (KOS-ADLS) Scale | At 6 months after intervention.
  The ADLS is a 14 item scale that queries patients about how their knee symptoms effect their ability to perform general daily activities (6 items) as well as how their knee condition effects their ability to perform specific functional tasks (8 items). Each item is scored 0-5 with 5 indicating "no difficulty" and 0 representing "unable to perform". The highest possible score is 70. The scores of all items are summed, divided by 70, then multiplied by 100 to give an overall ADLS percent rating. Higher percentages reflect higher levels of functional ability. This scale would be appropriate for patients who either do not participate in sports or recreational activities or for those who have not yet progressed to performing these activities
Knee Outcome Survey Activities of Daily Living (KOS-ADLS) Scale | At 12 months after intervention.
  The ADLS is a 14 item scale that queries patients about how their knee symptoms effect their ability to perform general daily activities (6 items) as well as how their knee condition effects their ability to perform specific functional tasks (8 items). Each item is scored 0-5 with 5 indicating "no difficulty" and 0 representing "unable to perform". The highest possible score is 70. The scores of all items are summed, divided by 70, then multiplied by 100 to give an overall ADLS percent rating. Higher percentages reflect higher levels of functional ability. This scale would be appropriate for patients who either do not participate in sports or recreational activities or for those who have not yet progressed to performing these activities
Knee Outcome Survey Activities of Daily Living (KOS-ADLS) Scale | At 24 months after intervention.
  The ADLS is a 14 item scale that queries patients about how their knee symptoms effect their ability to perform general daily activities (6 items) as well as how their knee condition effects their ability to perform specific functional tasks (8 items). Each item is scored 0-5 with 5 indicating "no difficulty" and 0 representing "unable to perform". The highest possible score is 70. The scores of all items are summed, divided by 70, then multiplied by 100 to give an overall ADLS percent rating. Higher percentages reflect higher levels of functional ability. This scale would be appropriate for patients who either do not participate in sports or recreational activities or for those who have not yet progressed to performing these activities
Knee laxity | At 12 months after intervention.
  The side to side knee joint laxity of patients after anterior cruciate ligament surgery can be divided into four grades: grade A: -1~2mm(0+), grade B: 3~5mm (1+), grade C: 6~10mm (2+) and D Grade: >10mm(3+) assessed by Lachman test of physical examination.
Knee laxity | At 6 months after intervention.
  The side to side knee joint laxity of patients after anterior cruciate ligament surgery can be divided into four grades: grade A: -1~2mm(0+), grade B: 3~5mm (1+), grade C: 6~10mm (2+) and D Grade: >10mm(3+) assessed by Lachman test of physical examination.
Quadriceps strength | At 6 months after intervention.
  Side to side quadriceps strength assessed by Biodex arthrometer test
Quadriceps strength | At 12 months after intervention.
  Side to side quadriceps strength assessed by Biodex arthrometer test
Lysholm score | At 6 months after intervention.
  Patients will be asked to fill out the Lysholm score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Lysholm score | At 12 months after intervention.
  Patients will be asked to fill out the Lysholm score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Lysholm score | At 24 months after intervention.
  Patients will be asked to fill out the Lysholm score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | At 6 months after intervention.
  Patients will be asked to fill out the KOOS score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | At 12 months after intervention.
  Patients will be asked to fill out the KOOS score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | At 24 months after intervention.
  Patients will be asked to fill out the KOOS score to document the functional status. The minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Tegner Score | At 6 months after intervention.
  Patients will be asked to fill out the Tegner score to document the functional status. The minimum is 0 and the maximum value is 10. Higher scores mean a better outcome.
Tegner Score | At 12 months after intervention.
  Patients will be asked to fill out the Tegner score to document the functional status. The minimum is 0 and the maximum value is 10. Higher scores mean a better outcome.
Tegner Score | At 24 months after intervention.
  Patients will be asked to fill out the Tegner score to document the functional status. The minimum is 0 and the maximum value is 10. Higher scores mean a better outcome.
hort Form (SF)-36,The medical outcome study 36-items short form health survey (SF-36) | At 6 months after intervention.
  Patients will be asked to fill out the SF-36 to document the quality of life . General health-related quality of life: SF-36 physical component score (range 0 to 100; higher score = better health state) at 2 yearsTh minimum is 0 and the maximum value is 100. Higher scores mean a better outcome.
Magnetic resonance imaging (MRI) | At 6 months after intervention.
  Magnetic resonance imaging was used to compare lateral comparisons of ligament healing and ACL graft healing after conservative treatment, meniscal damage and knee cartilage damage after intervention.
Magnetic resonance imaging (MRI) | At 12 months after intervention.
  Magnetic resonance imaging was used to compare lateral comparisons of ligament healing and ACL graft healing after conservative treatment, meniscal damage and knee cartilage damage after intervention.
Knee laxity （KT-2000 arthrometer） | At 6 months after intervention.
  The knee laxity test of the forward KT-2000 measured knee laxity at pressures of 132Nt, 88Nt, 66Nt, and 44Nt, respectively, while the back-pushing KT-2000 was measured at -132NT, 88Nt, 66Nt, and -44Nt. The foward-pushing KT-2000 asessed side-to-side can be stratified into five levels are (A) < - 1 mm, (B) - 1 to 1 mm, (C) 1-3 mm, (D) 3-5 mm and (E) > 5 mm.
  The back-pushing KT-2000 is also divided into side to side differences as (A) < - 2 mm, (B) - 2 to - 0.5 mm, (C) - 0.5 to 0.5 mm, (D) 0.5-1 mm and ( E) > 1 mm.
Knee laxity （KT-2000 arthrometer） | At 12 months after intervention.
  The knee laxity test of the forward KT-2000 measured knee laxity at pressures of 132Nt, 88Nt, 66Nt, and 44Nt, respectively, while the back-pushing KT-2000 was measured at -132NT, 88Nt, 66Nt, and -44Nt. The foward-pushing KT-2000 asessed side-to-side can be stratified into five levels are (A) < - 1 mm, (B) - 1 to 1 mm, (C) 1-3 mm, (D) 3-5 mm and (E) > 5 mm.
  The back-pushing KT-2000 is also divided into side to side differences as (A) < - 2 mm, (B) - 2 to - 0.5 mm, (C) - 0.5 to 0.5 mm, (D) 0.5-1 mm and ( E) > 1 mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anderson AF, Irrgang JJ, Kocher MS, Mann BJ, Harrast JJ; International Knee Documentation Committee. The International Knee Documentation Committee Subjective Knee Evaluation Form: normative data. Am J Sports Med. 2006 Jan;34(1):128-35. doi: 10.1177/0363546505280214. Epub 2005 Oct 11. PMID 16219941